CLINICAL TRIAL: NCT04068012
Title: A Computerized Decision Support Tool for Ventilator Management in Pediatric Acute Respiratory Distress Syndrome Pilot Study
Brief Title: Clinical Decision Support Tool in PARDS Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Christopher J. L. Newth, MD, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-19-00085
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Ventilation Therapy; Complications; Ventilator-Induced Lung Injury; Ards
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Ventilator management using the proposed protocol in both acute and weaning phases
  Interventions: Other: Ventilator protocol

INTERVENTIONS:
Other: Ventilator protocol — open loop ventilator management by a computer based protocol

SUMMARY:
Previous clinical trials in adults with acute respiratory distress syndrome (ARDS) have demonstrated that ventilator management choices can improve Intensive Care Unit (ICU) mortality and shorten time on mechanical ventilation. This study seeks to scale an established Clinical Decision Support (CDS) tool to facilitate dissemination and implementation of evidence-based research in mechanical ventilation of infants and children with pediatric ARDS (PARDS).

This will be accomplished by using CDS tools developed and deployed in Children's Hospital Los Angeles (CHLA) which are based on the best available pediatric evidence, and are currently being used in an NHLBI funded single center randomized controlled trial (NCT03266016, PI: Khemani). Without CDS, there is significant variability in ventilator management of PARDS patients both between and within Pediatric ICUs (PICUs), but clinicians are willing to accept CDS recommendations. The CDS tool will be deployed in multiple PICUs, targeting enrollment of up to 180 children with PARDS. Study hypotheses:

1. The CDS tool in will be implementable in nearly all participating sites
2. There will be > 80% compliance with CDS recommendations and
3. The investigators can implement automatic data capture and entry in many of the ICUs

Once feasibility of this CDS tool is demonstrated, a multi-center validation study will be designed, which seeks to determine whether the CDS can result in a significant reduction in length of mechanical ventilation (LMV).

DETAILED DESCRIPTION:
The central hypothesis is that CDS will help standardize ventilator management consistent with evidence-based recommendations leading to shorter LMV by limiting VILI (Ventilator Induced Lung Injury), preventing VIDD (Ventilator Induced Diaphragm Dysfunction) and allowing earlier recognition that patients are ready for liberation from the ventilator. However, key questions must be addressed prior to wide dissemination of this CDS tool:

Specific Aim 1: To assess the feasibility of implementing a web-based, de-identified CDS tool for MV in pediatric ARDS in multiple PICUs. Hypothesis: this CDS tool will be implementable in all PICUs to function consistent with each hospital's specific Information Technology (IT) capabilities.

Specific Aim 2: To assess the acceptability and compliance with recommendations from the CDS tool related to oxygenation, ventilation, weaning and extubation readiness testing in PARDS patients at each of the participating PICUs (anticipated 20 patients enrolled per site). Hypothesis: over time, adherence with recommendations in each of these domains will exceed 80% in all PICUs.

Specific Aim 3: To implement methods for automated data capture within CDS to provide the right information, to the right person, using the right format, in the right channel and at the right time during workflow ("CDS Five Rights") framework, which can be adapted to the individual IT capabilities at each hospital. Hypothesis: Over 90% of necessary data can be pulled into the CDS in an automated fashion in sites which have access to electronic data capture of ventilator settings and blood gases.

Patients will be managed on the eVentilator protocol (the CDS tool), through the acute, stable and weaning phases of mechanical ventilation, including Spontaneous Breathing tests (SBTs) and Extubation Readiness tests.

Data will be qualitatively assessed for implementation barriers. Acceptance and rejection and mode stratification will be examined. Data needed for the CDS protocol will be available electronically or can be interfaced through the bedside monitor.

Patients will be on the CDS protocol, as intent to treat, while patient is on invasive mechanical ventilation, capped at 28 days, limitation of care, or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Children > 1 month of age and >44 weeks gestation and ≤ 18 years of age AND
* Supported on mechanical ventilation with pulmonary parenchymal disease (i.e. Pediatric Acute Respiratory Distress Syndrome (PARDS)) with Oxygen Saturation Index (OSI) ≥ 5) or Oxygenation Index (OI) ≥ 4 AND
* Who are within 72 hours of initiation of invasive mechanical ventilation AND
* Who are anticipated to require >72 hours mechanical ventilation.

Exclusion Criteria:

* Conditions on enrollment that preclude conventional methods of weaning (i.e., status asthmaticus, severe lower airway obstruction, bronchiolitis, critical airway, Extra Corporeal Life Support (ECLS), intubation for Upper Airway Obstruction, Do Not Resuscitate orders, severe chronic respiratory failure, spinal cord injury above lumbar region, cyanotic heart disease (unrepaired or palliated)) OR
* Conditions precluding the use of permissive hypercapnia or hypoxemia (i.e. intracranial hypertension, severe pulmonary hypertension)
* Primary Attending physician refuses to enroll the patient

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Implementation Feasibility | through study completion - each patient will be capped at 28 days, limitation of care, or death, whichever comes first.
  The main outcome for Aim 1 is the ability to install the CDS tool in at least 7 of the 9 potential institutions and get data from each of the minimum of 140 patients anticipated to be enrolled. The survey data will be qualitatively assessed for themes related to barriers to implementation and consider this in future refinements of the CDS tool.
Aim 2: Protocol Adherence | through study completion - each patient will be capped at 28 days, limitation of care, or death, whichever comes first.
  Acceptance of recommendations (between 75-85%) will be the main outcome used to determine correctness of interpretation and acceptability of the CDS Tool.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Newth, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (8):
- United States (6):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Penn State University, Hershey, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- CHU Sainte-Justine, Montreal, Quebec, Canada
- Ospedale Pediatrico Bambino Gesu, Roma, Italy

REFERENCES:
- [Background] Hotz JC, Bornstein D, Kohler K, Smith E, Suresh A, Klein M, Bhalla A, Newth CJ, Khemani RG. Real-Time Effort Driven Ventilator Management: A Pilot Study. Pediatr Crit Care Med. 2020 Nov;21(11):933-940. doi: 10.1097/PCC.0000000000002556. PMID 32976348
- [Background] Khemani RG, Hotz JC, Klein MJ, Kwok J, Park C, Lane C, Smith E, Kohler K, Suresh A, Bornstein D, Elkunovich M, Ross PA, Deakers T, Beltramo F, Nelson L, Shah S, Bhalla A, Curley MAQ, Newth CJL. A Phase II randomized controlled trial for lung and diaphragm protective ventilation (Real-time Effort Driven VENTilator management). Contemp Clin Trials. 2020 Jan;88:105893. doi: 10.1016/j.cct.2019.105893. Epub 2019 Nov 16. PMID 31740425